CLINICAL TRIAL: NCT04729257
Title: Norms Expansion and Validation for IntelliSpace Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Collaborators: Research America Inc. (Industry); Qserve (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ICBE-S-000233
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Cognitive Functioning of Healthy Individuals
Keywords: Cognitive model; Cognitive assessment; Digital cognitive tests; Automated scoring; Algorithms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (6):
- Group A1 (Norms + Validation, 18-49 years) + Group A2 (Validation, 50+ years) (Other): Visit 1: Participants' cognition is measured using digital tests. Visit 2: Participants' cognition is measured using paper-pencil tests.
  Interventions: Device: Philips IntelliSpace Cognition (ISC).; Diagnostic Test: Paper-Pencil Tests.
- Group B (Validation, 18+) (Other): Visit 1: Participants' cognition is measured using paper-pencil tests. Visit 2: Participants' cognition is measured using digital tests.
  Interventions: Device: Philips IntelliSpace Cognition (ISC).; Diagnostic Test: Paper-Pencil Tests.
- Group C1 (Norms + Validation, 18-49 years) + Group C2 (Validation, 50+ years) (Other): Visit 1: Participants' cognition is measured using digital tests. Visit 2: Participants' cognition is measured using digital tests.
  Interventions: Device: Philips IntelliSpace Cognition (ISC).
- Group D (Validation, 18+) (Other): Visit 1: Participants' cognition is measured using paper-pencil tests. Visit 2: Participants' cognition is measured using paper-pencil tests.
  Interventions: Diagnostic Test: Paper-Pencil Tests.
- Group E (Norms, 18-49 years) (Other): Visit 1: Participants' cognition is measured using digital tests. Visit 2: N/A
  Interventions: Device: Philips IntelliSpace Cognition (ISC).
- Group F (Norms, 80-95 years) (Other): Visit 1: Participants' cognition is measured using digital tests. Visit 2: N/A
  Interventions: Device: Philips IntelliSpace Cognition (ISC).

INTERVENTIONS:
Device: Philips IntelliSpace Cognition (ISC). — Philips ISC is a Class-II Medical Device in the US that aids in assessing cognition and helps inform the HealthCare Professional (HCP) to make a diagnosis and treatment plan. ISC can be used in a variety of healthcare environments such as neurology and neuropsychology practices.
  Arms: Group A1 (Norms + Validation, 18-49 years) + Group A2 (Validation, 50+ years); Group B (Validation, 18+); Group C1 (Norms + Validation, 18-49 years) + Group C2 (Validation, 50+ years); Group E (Norms, 18-49 years); Group F (Norms, 80-95 years)
Diagnostic Test: Paper-Pencil Tests. — The same cognitive tests that are on the ISC platform are performed using paper and pencil (rather than digitally) as is the case in standard clinical practice.
  Arms: Group A1 (Norms + Validation, 18-49 years) + Group A2 (Validation, 50+ years); Group B (Validation, 18+); Group D (Validation, 18+)

SUMMARY:
This study aims to expand the normative dataset for Philips IntelliSpace Cognition to include ages 18-49 and 80+ and aims to validate two new digital tests.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 years or older.
* Participant's primary language (language most often spoken) must be American English.
* Participant is able to see well (naturally or corrected by means of eyeglasses or lenses).
* Participant is able to hear well (naturally of corrected by means of a hearing aid).
* Participant is able to use their fingers, hands and arms to write symbols.
* Participant has valid health insurance in USA.
* Participant is able to give informed consent.
* Participant is able to understand test instructions and participate fully in testing.
* Participant has normal fine and gross motor ability.

Exclusion Criteria:

Inclusion Criteria:

* Participant is 18 years or older.
* Participant's primary language (language most often spoken) must be American English.
* Participant is able to see well (naturally or corrected by means of eyeglasses or lenses).
* Participant is able to hear well (naturally of corrected by means of a hearing aid).
* Participant is able to use their fingers, hands and arms to write symbols.
* Participant has valid health insurance in USA.
* Participant is able to give informed consent.
* Participant is able to understand test instructions and participate fully in testing.
* Participant has normal fine and gross motor ability.

Exclusion Criteria:

* Participant is currently admitted to a hospital, assisted living, nursing home or a psychiatric facility.
* Participant is diagnosed with a neurological disorder or disease that may affect cognitive functioning (e.g., Parkinson's, brain tumor, stroke, Traumatic Brain Injury (TBI), epilepsy [if # seizures ≤ 2 and not receiving ongoing treatment for seizures, and not currently seeking medical evaluation or attention related to seizures, participant can be accepted], encephalitis, dementia).
* Participant is diagnosed with a language disorder or aphasia (expressive or mixed receptive/expressive) [if articulation disorder, participant can be accepted].
* Participant is diagnosed with a learning disorder.
* Participant is diagnosed with an autoimmune disorder that may affect cognitive functioning (e.g., LUPUS, Multiple Sclerosis).
* Participant is or was diagnosed with a current or past psychotic disorder (e.g., schizophrenia).
* Participant is diagnosed with a severe mood disorder [if Major Depressive Disorder in remission or with no current episode or Dysthymic Disorder or Adjustment Disorder, participant can be accepted].
* Participant is diagnosed with a severe anxiety disorder [if Phobia or Anxiety disorders with symptoms not significant enough to interfere with test performance, participant can be accepted].
* Participant is or was diagnosed with current or past Autism Spectrum Disorder or Intellectual Disability.
* Participant is diagnosed with a current substance abuse or dependence [if in remission ≥ 1 year, participant can be accepted].
* Participant has carried a substance abuse or dependence diagnosis for more than 10 years at any point in their life.
* Participant has an average alcohol consumption of 4 or more units per day.
* Participant uses medical marijuana.
* Participant uses recreational marijuana more than once a week.
* Participant uses recreational drugs other than alcohol and marijuana in the last 6 months (e.g., cocaine, ecstasy, LSD).
* Participant has been unconscious related to traumatic brain injury or 'medical condition' for more than 20 minutes [if medication-induced or due to heat stroke, participant can be accepted].
* Participant has stayed in a hospital overnight due to a head injury.
* Participant has had a medical event requiring resuscitation in which they were non-responsive for more than 15 minutes.
* Participant has received chemotherapy treatment in the past 2 months.
* Participant has received electroconvulsive therapy (ECT).
* Participant has received radiation to the central nervous system.
* Participant experiences a physical condition or illness that interferes with normal cognitive functioning at work, school, Instrumental Activities of Daily Living (IADLs) etc. [if diabetes or hypothyroidism or hypertension and if controlled, participant can be accepted].
* Participant is currently taking anti-convulsants (Depakote, Lamictal or Lyrica, Gabapentin, Keppra, Topamax, Divalproex Sodium, Valproate Sodium, Levetiracetam, Lamotrigine, Pregabalin, Topiramate).
* Participant is currently taking anti-psychotics (Abilify, Rexulti, Zyprexa, Clozaril, Clozapine, Latuda, Seroquel, Risperdal, Risperidone, Aripipazle, Bexipiprazole, Olanzapine, Lurasidone HCL, Quetiapine).
* Participant is currently taking benzodiazepines (Diazepams, Valium, Klonopin, Ativan, Xanax, Lorazepam, Alprazolam, Clonazepam).
* Participant is currently taking psychostimulants (Amphetamines, Adderall, Ritalin, Methamphetamines, Dextroamphetamine, Methylphenidate HCL). [if coffee, participant can be accepted].
* Participant is currently taking opioids (Oxycontin, Tramadol, Codeine, Dilaudid, Suboxone, Oxycodone, Percocet, Buprenorhine, Naloxone).
* Participant is currently taking antidepressants (Amitriptyline, Elavil, Pamelor, Tofranil, Vivactil, Imipramine, Protriptyline HCL). [if antidepressant that are not tricyclic, participant can be accepted].
* Participant is currently taking oxybutynin (Ditropan).
* Participant is currently seeking medical diagnostic procedures for cognitive difficulties from a medical professional.
* Participant has received neuropsychological testing before. [if previous MMSE(-2) or MoCA testing more than 6 months prior, participant can be accepted].
* Participant shows evidence of current cognitive impairment.
* Participant displays disruptive behavior or insufficient compliance with testing to ensure a valid assessment.
* Participant is primarily nonverbal or uncommunicative.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
1. Scores digital (ISC) tests [Time Frame: 1.5 hours]. Scores retrieved from all cognitive tests on the ISC platform. | 1.5 hours
or 1.5 hours]. Scores retrieved from Symbol Digit Modalities Test (SDMT) + Naming Test (NT) or all paper-based cognitive tests | 0.75 h or 1.5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Research America Inc., Newtown Square, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No